CLINICAL TRIAL: NCT05192486
Title: An Open-Label, Multi-Center, Phase Ib/II Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of Tetra-specific Antibody GNC-038 in Participants With Recurrent or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Study of GNC-038, a Tetra-specific Antibody, in Participants With R/R Diffuse Large B-cell Lymphoma (DLBCL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-102
Record Dates: First submitted 2021-12-15; First posted 2022-01-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-038 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-038

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion

SUMMARY:
In this study, the safety and preliminary efficacy of GNC-038 in participants with recurrent or refractory Diffuse Large B-cell lymphoma (DLBCL) will be investigated to assess the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MAD) for MTD is not reached of GNC-038. The recommended dose for phase II (RP2D) clinical study will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. he participants could understand and sign the informed consent form, and must participate voluntarily;
2. No gender limit;
3. Age: ≥18 years old and ≤75 years;
4. Expected survival time ≥ 3 months;
5. Has suffered from Diffuse Large B-cell lymphoma (DLBCL) confirmed by histology or cytology;
6. a. Those who have recurrent or refractory Diffuse Large B-cell lymphoma (DLBCL).

   b. Recurrent or refractory participants that are, determined by the investigators, not applicable/tolerated to other treatments.

   Recurrent and refractory are defined as follows:

   Recurrent is the progression of disease after adequate treatment to remission, with at least one regimen containing rituximab.

   Refractory refers to failure to respond to adequate treatment with rituximab containing regimen (combination chemotherapy or monotherapy) or disease progression during treatment/within 6 months of completion of adequate treatment.

   "Adequate treatment with rituximab regimen" refers to the completion of rituximab combined with chemotherapy based on pathological type and disease stage requirements, or rituximab monotherapy with 375 mg/m2 injections at least 4 times a week. "Progress during treatment" requires completion of at least one cycle of rituximab plus chemotherapy or monotherapy if progress during induction therapy; At least one injection is completed if progress is made during maintenance therapy. "Mitigation" includes complete and partial mitigation.
7. There are measurable lesions during the screening period (any long diameter of lymph node lesions ≥ 1.5 cm or any long diameter of extra-nodal lesions greater than 1.0 cm);
8. Physical fitness score ECOG≤2；
9. The toxicity of the previous anti-tumor therapy has been restored to the level ≤1 defined by NCI-CTCAE v5.0 (the investigators considered indicators that might be associated with the disease, such as anemia, and excluded toxicities that the investigators considered to be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy);
10. The organ function within 7 days prior to the first administration meets the following requirements:

    * Bone marrow function: In the case of no blood transfusion, no use of G-CSF (no use of long-acting whitening needles within 2 weeks) and drug correction within 7 days prior to screening, the absolute value of neutrophil count (ANC) ≥1.0×109/L (participants with bone marrow infiltration ≥0.5×109/L); Hemoglobin ≥80 g/L (for participants with bone marrow infiltration, ≥70 g/L); Platelet count ≥50×109/L;
    * Liver function: In the absence of hepatoprotective drugs for correction within 7 days prior to screening, total bilirubin (TBIL) ≤ 1.5 ULN (TBIL ≤3 ULN in participants with Gilbert's syndrome), transaminase (AST/ALT) ≤ 2.5 ULN (participants with tumor infiltration in the liver ≤5.0 ULN);
    * Kidney function: creatinine (Cr) ≤ 1.5 ULN and creatinine clearance (Ccr) ≥ 50 mL/min (according to the Cockcroft and Gault formula);
    * Routine urine / 24h urine protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24h urine protein < 1g can be included);
    * Cardiac function: left ventricular ejection fraction ≥50%;
    * Coagulation function: fibrinogen (FIB) ≥1.5g/L; activated partial thromboplastin time (APTT) ≤1.5×ULN; prothrombin time (PT) ≤1.5×ULN.
11. Female participants with fertility or male participants whose partner(s) are fertile must take effective contraceptive measures from 7 days prior to the first administration to 24 weeks after the administration. Female participants with fertility must have a negative serum/urine pregnancy test in 7 days prior to the first dose.
12. The subjects are able and willing to follow the visits, treatment plans, laboratory tests, and other study-related procedures specified in the study protocol.

Exclusion Criteria:

1. Has grade 3 or above lung disease defined according to NCI-CTCAE v5.0; Patients with current interstitial lung disease (ILD) (except those who have recovered from previous interstitial pneumonia;
2. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc;
3. Active tuberculosis;
4. Participants at risk of active autoimmune diseases, such as: systemic lupus erythematosus, systemic treatment of psoriasis, rheumatoid arthritis, inflammatory bowel disease, and hashimoto's thyroiditis, etc., with the exception of type I diabetes, only replacement therapy can control the hypothyroidism, no systemic treatment of skin disease (such as vitiligo, psoriasis), B cells caused by autoimmune disease;
5. Complicated with other malignant tumors within 5 years prior to GNC-038 treatment, except for non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ, gastrointestinal intramucosal cancer, breast cancer and localized prostate cancer that have been cured and have not recurred within 5 years;
6. HBsAg or HBcAb positive and HBV-DNA test ≥ULN; HCV antibody positive and HCV-RNA≥ULN; HIV antibody positive;
7. Participants with poorly controlled hypertension by antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg);
8. History of severe heart disease, including but not limited to:

   * There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias, III grade atrioventricular block, which require clinical intervention;
   * Participants with prolonged QT interval (male QTc > 450 msec or female QTc > 470 msec);
   * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months before the first administration;
   * New York Heart Association (NYHA) grade II, III or IV congestive heart failure;
9. Patients with a history of allergy to recombinant humanized antibodies or to any excipient component of GNC-038;
10. Pregnant or breastfeeding women;
11. There is an invasion of the central nervous system;
12. Has undergone major surgery within 28 days prior to the administration of this study, or planned to undergo major surgery during the study period (except for surgery such as puncture or lymph node biopsy);
13. Has accepted organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLo-HSCT);
14. Has accepted autologous hematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks prior to GNC-038 treatment;
15. Currently using immunosuppressive agents within 2 weeks prior to GNC-038 treatment, including but not limited to: Cyclosporine, tacrolimus, etc.; receiving high-dose glucocorticoids within 2 weeks prior to GNC-038 treatment (longer than 14 days, a stable dose of >30 mg of prednisone or other glucocorticoids at the same dose per day);
16. Has received radiotherapy within 4 weeks prior to GNC-038 treatment;
17. Has received anti-CD20 or anti-CD79b treatment within 4 weeks prior to GNC-038 treatment, and continued to respond;
18. Has received chemotherapy, small molecule targeted drugs within 2 weeks prior to GNC-038 treatment;
19. Has received CAR-T treatment within 12 weeks prior to GNC-038 treatment.
20. Has participated in any other clinical trials within 4 weeks prior to GNC-038 treatment;
21. Other conditions that the investigator believes that it is not suitable for participating in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 21 days after the first dose of GNC-038
  The incidence and severity of adverse events during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Maximum tolerated dose (MTD) or maximum administrated dose (MAD) | Up to 21 days after the first dose of GNC-038
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
The recommended dose for phase II clinical study（RP2D） | Up to 21 days after the first dose of GNC-038
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.

SECONDARY OUTCOMES:
ORR (Objective Response Rate ) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
PFS (Progression-free Survival) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
DCR (Disease Control Rate) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
DOR (Duration of Response) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
CR (Complete Response) | Up to approximately 24 months
  Disappearance of all target lesions.
Adverse Events of special interest (AESI) | Up to approximately 24 months
  AESI is an event of scientific and medical interest specific to the sponsor's product or research project.
Peak Plasma Concentration（Cmax) | Up to 21 days after the first dose of GNC-038
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Incidence and titer of ADA (Anti-drug antibody) | Up to approximately 24 months
  Frequency and titer of anti-GNC-038 antibody (ADA) will be evaluated.
Incidence and titer of Nab | Up to approximately 24 months
  Incidence and titer of Nab of GNC-038 will be evaluated.
Trough steady-state concentration（Css） | Up to 14 days after the first dose of GNC-038
  Concentration of GNC-038 at steady state plateau will be investigated.
Time to reach maximum concentration (Tmax) | Up to 21 days after the first dose of GNC-038
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
AUC0-inf | Up to 21 days after the first dose of GNC-038
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite (AUC0-inf).
AUC0-t | Up to 21 days after the first dose of GNC-038
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC0-t).
Plasma clearance （CL） | Up to 21 days after the first dose of GNC-038
  To study the serum clearance rate of GNC-038 per unit time.
Elimination half life （T1/2） | Up to 21 days after the first dose of GNC-038
  Half-life (T1/2) of GNC-038 will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital
Locations (4):
- China (4):
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No